CLINICAL TRIAL: NCT00000976
Title: A Phase I Study of the Safety and Pharmacokinetics of Recombinant Human CD4-Immunoglobulin G (rCD4-IgG) Administered by Intravenous Bolus Injection in Combination With Oral Zidovudine in Patients With AIDS and AIDS-Related Complex
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Genentech, Inc. (Industry)
Purpose: Treatment
Other Study IDs: ACTG 134; D0156g
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2008-08-06 (Estimated); Status verified 1994-12

CONDITIONS: HIV Infections
Keywords: Recombinant Proteins; Injections, Intravenous; IgG; Drug Evaluation; Administration, Oral; Acquired Immunodeficiency Syndrome; Antigens, CD4; Zidovudine; Carrier Proteins
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — CD4 Immunoadhesins; Zidovudine

INTERVENTIONS:
Drug: CD4-IgG
Drug: Zidovudine

SUMMARY:
To determine the safety profile of recombinant human CD4-immunoglobulin G (CD4-IgG) and zidovudine (AZT) combination therapy in patients with AIDS or AIDS-related complex (ARC); to assess pharmacokinetic (blood level) properties of CD4-IgG in combination with AZT; and to obtain preliminary indication of the antiviral and immunologic effects of CD4-IgG in combination with AZT in patients with AIDS and ARC.

Treatment of AIDS has been directed toward the underlying retroviral infection as well as toward specific opportunistic infections and malignancies that are associated with the syndrome. The most extensively studied drugs are reverse transcriptase inhibitors such as AZT and other nucleoside analogs, including didanosine (ddI) and dideoxycytidine (ddC). The most extensive clinical experience has been achieved with AZT. These clinical trials indicated a decreased incidence of opportunistic infection and increased survival in patients with AIDS. However, AZT treatment is associated with dose-limiting toxicities. Additionally, identification of resistance to AZT has increased the need to test the effectiveness of AZT in combination with other drugs. CD4-IgG is capable of binding to HIV envelope protein (gp120) and inhibiting HIV infectivity in test tube studies. Potential therapeutic benefit in patients with HIV infection may be derived from CD4-IgG.

DETAILED DESCRIPTION:
Treatment of AIDS has been directed toward the underlying retroviral infection as well as toward specific opportunistic infections and malignancies that are associated with the syndrome. The most extensively studied drugs are reverse transcriptase inhibitors such as AZT and other nucleoside analogs, including didanosine (ddI) and dideoxycytidine (ddC). The most extensive clinical experience has been achieved with AZT. These clinical trials indicated a decreased incidence of opportunistic infection and increased survival in patients with AIDS. However, AZT treatment is associated with dose-limiting toxicities. Additionally, identification of resistance to AZT has increased the need to test the effectiveness of AZT in combination with other drugs. CD4-IgG is capable of binding to HIV envelope protein (gp120) and inhibiting HIV infectivity in test tube studies. Potential therapeutic benefit in patients with HIV infection may be derived from CD4-IgG.

AMENDED: Previously, rCD4-IgG had been administered on a mcg/kg basis. Subjects now receive rCD4-IgG as a fixed dose. Changes to the maintenance schedule were made to accommodate the new dosages. Original design: This study is divided into two parts: A pharmacokinetic evaluation, and a safety evaluation. The pharmacokinetic evaluation is done in selected patients. For the safety evaluation patients will receive rCD4-IgG at a fixed dose level twice weekly by intravenous bolus injection (over 1 minute) for 12 weeks. Zidovudine (AZT) is administered orally 3 times daily at one of two dose levels. Eight subjects, at least 4 of whom with p24 levels greater than 75 pg/m, are entered at each dose level of CD4-IgG beginning with dose level 1. If 3 or more patients at a dose level experience grade 3 or 4 toxicity then no further patients will be added to that or higher dose levels. Pharmacokinetics of CD4-IgG alone and in combination with AZT is evaluated in patients at dose level 2 only. Patients receive one IV bolus of CD4-IgG on day 1 and samples are drawn beginning 15-30 minutes prior to the CD4-IgG injection. There is an 8 day washout period. Beginning on day 9 and continuing through day 24, patients receive AZT daily. CD4-IgG is administered by IV bolus on day 16. Samples are drawn beginning 15-30 minutes prior to the injection of CD4-IgG. The pharmacokinetic evaluation terminates 8 days after the second CD4-IgG injection (day 24). Extended treatment will be made available to patients at the discretion of the Principal Investigator.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Topical acyclovir.

Patients must have the following:

* HIV seropositivity.
* Life expectancy of at least 3 months.
* No white or red blood cell casts in urine.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Serious active opportunistic infection or malignancies other than Kaposi's sarcoma.
* Kaposi's sarcoma requiring therapy, tumor-associated edema, or visceral disease.

Concurrent Medication:

Excluded:

* Intravenous acyclovir for Herpes.
* Interferon.
* Systemic corticosteroids.
* Nonsteroidal anti-inflammatory agents.
* Intravenous acyclovir.
* Other known immunomodulatory agents.
* Dideoxycytosine (ddC), didanosine (ddI).
* Other nucleoside analogs not specifically allowed.
* Other experimental therapy.

Patients with the following are excluded:

* Serious active opportunistic infection or malignancies other than Kaposi's sarcoma.
* More than 120 days (total) of prior zidovudine (AZT) therapy.
* Currently receiving intravenous acyclovir for Herpes.

Prior Medication:

Excluded:

* > 120 days total of prior zidovudine (AZT) therapy.
* Excluded within 3 weeks of study entry:
* Immunomodulatory agents.
* Other experimental therapy.

Prior Treatment:

Excluded within the past 3 months:

* Transfusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40

CONTACTS AND LOCATIONS:
Overall Officials: D Richman, Study Chair; M Fischl, Study Chair
Locations (3):
- United States (3):
  - Univ of California / San Diego Treatment Ctr, San Diego, California
  - Univ of Miami School of Medicine, Miami, Florida
  - Univ of Massachusetts, Worcester, Massachusetts

REFERENCES:
- [Background] Meng TC, Fischl MA, Cheeseman SH, Spector SA, Resnick L, Boota A, Petrakis T, Wright B, Richman DD. Combination therapy with recombinant human soluble CD4-immunoglobulin G and zidovudine in patients with HIV infection: a phase I study. J Acquir Immune Defic Syndr Hum Retrovirol. 1995 Feb 1;8(2):152-60. PMID 7834398